CLINICAL TRIAL: NCT00674739
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multi-center, Efficacy and Safety Study of Imiquimod Creams in the Treatment of External Genital Warts
Brief Title: Safety and Effectiveness Study of Imiquimod Creams in the Treatment of External Genital Warts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Jason Wu, MD / Exective Director, Product Development, Graceway Pharmaceuticals, LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GW01-0801
Record Dates: First submitted 2008-05-07; First posted 2008-05-08 (Estimated); Results first posted 2011-05-18 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Genital Warts
Keywords: external genital warts; perianal warts; condylomata acuminata; venereal warts; HPV types 6 and 11
MeSH Terms: conditions — Condylomata Acuminata | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- imiquimod cream (Experimental): 2.5% imiquimod cream applied daily to wart area for up to 8 weeks
  Interventions: Drug: Imiquimod
- 3.75% imiquimod cream (Experimental): 3.75% imiquimod cream applied daily to wart areas for up to 8 weeks.
  Interventions: Drug: 3.75% imiquimod cream
- placebo cream (Placebo Comparator): placebo cream applied daily to wart areas for up to 8 weeks
  Interventions: Drug: placebo cream

INTERVENTIONS:
Drug: Imiquimod — daily topical application for up to 8 weeks
  Other Names: imiquimod 2.5% topical creram
  Arms: imiquimod cream
Drug: 3.75% imiquimod cream — 3.75% imiquimod cream applied daily to wart areas for up to 8 weeks.
  Other Names: 3.75% imiquimod topical cream
  Arms: 3.75% imiquimod cream
Drug: placebo cream — placebo cream applied daily to wart areas for up to 8 weeks
  Other Names: placebo matching cream
  Arms: placebo cream

SUMMARY:
The purpose of this study is to determine whether imiquimod creams are effective in treating external genital warts (EGW). The secondary objective of this study is to provide information on recurrence of EGW. Additionally the study will also look at any adverse events associated with the use of the creams.

External genital and perianal warts are caused by the infection of human papillomavirus or HPV. HPV infection is a sexually transmitted disease (STD). External genital warts look like small flesh-colored, pink, or red growths on or around the external skin of sex organs or perianal area. The warts may look similar to the small parts of a cauliflower or they may be very tiny and difficult to see. They often appear in clusters of three or four, and may grow and spread rapidly. They usually are not painful, although they may cause mild pain, bleeding, and itching.

ELIGIBILITY:
Inclusion Criteria:

* In good general health
* Diagnosis of external genital / perianal warts with at least 2 warts and no more than 30 warts
* Negative pregnancy test (for women who are able to become pregnant)

Exclusion Criteria:

* Women who are pregnant, lactating or planning to become pregnant during the study
* Evidence of clinically significant or unstable disease (such as stroke, heart attack)
* Have any of the following conditions: HIV infection; current or history of high risk HPV infection (e.g., HPV 16, 18, etc.); outbreak of herpes genitalia in the wart areas; internal warts requiring or undergoing treatment; dermatological disease (e.g., psoriasis) or skin condition in the wart areas
* Have received specific treatments in the treatment area(s) within the designated time period prior to study treatment initiation.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, MD, Study Director — Graceway Pharmaceuticals
Locations (30):
- United States (30):
  - WILMAX Clinical Research, Mobile, Alabama
  - Montgomery Women's Health Associates, Montgomery, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Premier Pharmaceutical Research, Tempe, Arizona
  - Visions Clinical Research, Tucson, Arizona
  - Edinger Medical Group Clinical Research Center, Fountain Valley, California
  - East Bay Dermatology Medical Group, Fremont, California
  - Coastal Medical Research Group, San Luis Obispo, California
  - Torrance Clinical Research, Torrance, California
  - Clinicos, LLC, Colorado Springs, Colorado
  - Colorado Medical Research Center, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Miami Research Associates, South Miami, Florida
  - Discovery Clinical Research, Sunrise, Florida
  - Perimeter Institute for Clinical Research, Atlanta, Georgia
  - Medical College of Georgia, Augusta, Georgia
  - Atlanta North Gynecology, Roswell, Georgia
  - Indiana University Infectious Disease Research Group, Indianapolis, Indiana
  - Dermatology Practice, Ann Arbor, Michigan
  - Alegent Health Clinic, Omaha, Nebraska
  - Private Practice, Great Neck, New York
  - Private Practice, Purchase, New York
  - State University of NY Stony Brook, Stony Brook, New York
  - Philadelphia Institute of Dermatology, Philadelphia, Pennsylvania
  - Professional Quality Research, Women Partners in Health, Austin, Texas
  - Professional Quality Research, The Urology Team, Austin, Texas
  - University of Texas Southwestern Medical Center Dermatology Dept, Dallas, Texas
  - Progressive Clinical Research, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from June to December 2008 from 30 clinical study centers in the USA
Groups:
- 2.5% Imiquimod Cream: 2.5% imiquimod cream applied once daily to wart areas for up to 8 weeks
- 3.75% Imiquimod Cream: 3.75% imiquimod cream applied once daily to wart areas for up to 8 weeks
- Placebo: Placebo cream applied once daily to wart areas for up to 8 weeks
Period: Overall Study
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Started | 178 | 195 | 97
Completed | 121 | 136 | 65
Not Completed | 57 | 59 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo | Total
Number analyzed (Participants) | 178 | 195 | 97 | 470
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 3 | 4 | 11
  Between 18 and 65 years | 173 | 189 | 91 | 453
  >=65 years | 1 | 3 | 2 | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 32.7 (11.3) | 32.5 (11.6) | 30.5 (10.6) | 32.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 100 | 50 | 245
  Male | 83 | 95 | 47 | 225
Region of Enrollment [Number; unit: participants]
  United States | 178 | 195 | 97 | 470

OUTCOME MEASURES:

1. Secondary Outcome: Safety Variables Include Adverse Reactions (AEs), Local Skin Reactions (LSRs), and Number of Subjects Who Took Rest Periods During the Treatment Period.
Description: Local skin reactions in the treatment and/or immediate surrounding area were clinically identified as: erythema, edema, weeping/exudate, flaking/scaling/dryness, and erosion/ulceration. LSRs were visually assessed by investigator at each visit.
  Rest period was a temporary interruption of dosing dur to intolerable LSRs.
Time Frame: Up to 16 weeks
Measure: Number; unit: participants
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Number analyzed (Participants) | 178 | 195 | 97
participants
  Adverse Reactions | 27 | 30 | 2
  Local Skin Reactions | 110 | 144 | 29
  Number of Subjects with Rest Period in Treatment | 49 | 59 | 1

2. Primary Outcome: Proportion of Subjects With Complete Clearance of All Warts (Both Presented at Baseline and Newly Emerged Warts) at End of Study
Description: Proportion of subjects with complete clearance of all warts (both presented at Baseline and newly emerged warts) at End of Study. Primary analysis performed on the Intent to Treat population with imputation (Last Observation Carried Forward)for missing data points.
Time Frame: Up to 16 weeks
Population: Intention to treat
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Number analyzed (Participants) | 178 | 195 | 97
participants | 0.191 [0.136 to 0.257] | 0.272 [0.211 to 0.340] | 0.103 [0.051 to 0.181]

3. Secondary Outcome: Treatment Related Adverse Events
Description: Numbers of subjects in each treatment group reporting one or more adverse events
Time Frame: Up to 16 weeks
Population: Patients with adverse events considered probably related or related to the administration of the product.
Measure: Number; unit: Participants
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Number analyzed (Participants) | 178 | 195 | 97
Participants | 27 | 30 | 2

ADVERSE EVENTS:
Time Frame: One year
Description: The study duration included 5 month enrollment period, up to 28 week of study period, so total duration from first patient enrolled to the last patient completed study was approximately 12 months
Arm/Group | 2.5% Imiquimod Cream | 3.75% Imiquimod Cream | Placebo
Serious Adverse Events (participants affected / at risk) | 2/178 | 2/195 | 0/97
Other Adverse Events (participants affected / at risk) | 17/178 | 23/195 | 2/197
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.5% Imiquimod Cream (N=178) | 3.75% Imiquimod Cream (N=195) | Placebo (N=97)
Pelvic Mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Acute Surgical Abdomen
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) — Cholecystolithiasis
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) — Worsened iron deficiency anemia
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Worsening migraine headache
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Syncope
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2.5% Imiquimod Cream (N=178) | 3.75% Imiquimod Cream (N=195) | Placebo (N=197)
Application site pain (Skin and subcutaneous tissue disorders) | 12 (12) | 11 (11) | 1/97 (1)
Application site irritation (Skin and subcutaneous tissue disorders) | 5 (5) | 12 (12) | 1/97 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For few PIs, there were a restrict that the PI can not publish their trial results with 12 months from the completion of the trial.